CLINICAL TRIAL: NCT02180932
Title: Towards a Viral Etiology of Periodontal Disease in Relation to Radiotherapy Treatment of Head and Neck Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-GIRCI-01
Record Dates: First submitted 2014-05-20; First posted 2014-07-03 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2014-05

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- periodontal disease (Experimental): Saliva samples
  Interventions: Biological: periodontal pocket samples

INTERVENTIONS:
Biological: periodontal pocket samples

SUMMARY:
The treatment of otolaryngology (OLR) cancer is based on surgery, radiation, sometimes used in combination with chemotherapy. Patients treated with radiotherapy have multiple oral diseases: mucositis, hyposalivation, tissue fibrosis, exacerbation of periodontitis. Over 70% of patients with head and neck cancers treated with radiotherapy have a lower level of dental clinical attachment and 92% have loose teeth or missing. The management of these oral complications is a priority in OLR oncology. The aim is to improve the oral health of patients to achieve a comfortable life acceptable and necessary for healing.

This project proposes to deepen the investigation with two main objectives:

1. To study in vivo the effect of radiation treatment on the evolution of the viral flora of the periodontium in a cohort of patients and matched controls.
2. To study in vitro the effects of irradiation on the replication EBV (herpesvirus) in producing websites lymphoepithelial tonsillar, and atypical dendritic cells associated with EBV that existence were recently discovered.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients treated with curative radiotherapy on tumor site or surgery for cancer of the oral cavity and / or oropharynx
* Patients naive treatments for head and neck cancers
* Patients affiliated or beneficiary of a social security scheme
* Patients who gave informed consent in writing

Exclusion Criteria:

* Patients treated with neoadjuvant chemotherapy, adjuvant or concomitant
* Patients taking immunosuppressants after organ transplantation
* Taking anticoagulants incompatible with dental samples (possible bleeding)
* Patients edentulous and / or whose dental condition is incompatible with the dental samples

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Measure of level of EBV nucleic acids | day 1
Measure of level of EBV nucleic acids | day 180

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital saint Roch, Nice, France